CLINICAL TRIAL: NCT06706986
Title: ROSETTA- a Global Registry on Second GEneration and Long-acting InTegrase InhibiTor FAilures
Brief Title: A Global Registry on Second GEneration and Long-acting InTegrase InhibiTor FAilures
Acronym: ROSETTA
Status: Enrolling by invitation | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Luxembourg Institute of Health (Other Government); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Annemarie Wensing, Clinical Virologist, UMC Utrecht
Other Study IDs: V0002187
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: HIV; Therapy Failure
Keywords: integrase inhibitors; HIV drug resistance; subtype

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — If a center is not able to perform a genotypic resistance test, the ROSETTA team may isolate HIV DNA from a plasma sample to perform resistance testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Integrase strand transfer inhibitors (INSTI) inhibit HIV replication by preventing the integration of viral HIV DNA into the host's genome. INSTIs are used as part of combination antiretroviral therapy (cART) regimens for both treatment-naive and treatment experienced patients.

In clinical practice, virological failure to second generation INSTIs is rare and often without selection of known resistance mutations. Considering the use of INSTIs in first line regimens in high income countries and the increasing roll-out in lower and middle income countries, a better understanding of relevant resistance development and clinical failure is urgently needed.

The ROSETTA registry aims at systematically collecting otherwise scattered information on individual cases failing second generation integrase inhibitors, with the goal to inform policy and future use of INSTIs in the treatment of people living with HIV.

Attending physicians of individuals who are experiencing virological failure on a second generation integrase inhibitor-containing regimen are invited to contribute data to the registry.

DETAILED DESCRIPTION:
The ROSETTA study collects clinical data and HIV sequences from individuals experiencing failure of ART containing second generation INSTIs from Americas, Africa and Europe. If resistance testing is not available, the ROSETTA team can perform genotypic resistance testing of RT, protease, integrase and 3'-PPT.

Research objectives:

To set up a database with data of individuals who have experienced virological failure on a regimen containing a second generation INSTI To determine the prevalence of resistance mutations in integrase and 3'-PPT in the dataset To identify possible new resistance mutations outside integrase and 3'-PPT. providing additional funding is retrieved.

The study design will be a multicenter observational cohort study. Patients will be included from HIV care centers in Europe, America and Africa, if they fullfill the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection
* Using cART (any regimen) for at least the last 6 months
* Experiencing virological failure* on a second generation INSTI-containing regimen (including monotherapy and dual-therapy regimens)
* Data on current regimen and previous INSTI exposure available (start/stop dates and dosing mandatory)
* Integrase genotypic data available (performed locally) or a plasma/DBS (or CSF if available) sample(s) drawn at time of failure available to perform genotypic testing centrally * Virological failure is defined as at least 2 consecutive viral loads (VL) above 50 copies/mL in plasma or 1 VL above 200 copies/mL in plasma. We will also include patients who have a VL of >50 copies/mL in CSF, independent of the VL in plasma.

Exclusion Criteria:

* Submitted fasta file not passing quality control and unavailability of a stored sample to repeat sequence analysis
* Missing Mandatory data
* Documented treatment interruption for at least 2 weeks prior to viral load testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People living with HIV-1 experiencing virological failure to second-generation integrase inhibitors from Africa, Americas and Europe.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence and patterns of resistance in the dataset | 3 years
  The prevalence of resistance in the dataset in relation to HIV subtype and collected clinical parameters

SECONDARY OUTCOMES:
Identify new mutations related to integrase inhibitor resistance | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie MJ Wensing, MD,PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
ROSETTA will not own the data

REFERENCES:
- [Background] Special Issue: Abstract Supplement HIV Glasgow 10-13 November 2024, Glasgow, UK/Virtual. J Int AIDS Soc. 2024 Nov;27 Suppl 6(Suppl 6):e26370. doi: 10.1002/jia2.26370. No abstract available. PMID 39513741
- See also: Related Info — https://www.esar-society.eu/rosetta-registry/interest-in-rosetta-registry